CLINICAL TRIAL: NCT01406964
Title: Chlamidia Antibodies Test for Tubal Factor Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Juan Giles, IVI Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VLC-JD-0904-025
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Sterility
Keywords: Chlamidia Antibody test, Hysterosalpyngography, Tubal disease
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Arm A performs a CAT test to study tubal factor causes
  Interventions: Other: CAT test
- Arm B (Experimental): In Arm B a histerosalpingography is performed.
  Interventions: Other: Histerosalpingography

INTERVENTIONS:
Other: CAT test — A CAT test is performed in order to diagnose tubal factor causes
  Arms: Arm A
Other: Histerosalpingography — A Histerosalpingography is performed.
  Arms: Arm B

SUMMARY:
The aim of this study is to evaluate the usefulness of a Chlamydia Antibody Test for screening of tubal factor in patients who undergo artificial insemination.

ELIGIBILITY:
Inclusion Criteria:

* Age < 38 years
* FSH < 12.
* Treatment intrauterine insemination

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease
* Severe male factor
* Policystic ovarian syndrome
* Previous abdominal or uterine surgery
* Prevous abdominal or genital infections
* Uterine myomas
* Hidrosalpinx
* Uterine congenital abnormalities

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome using the two different treatments. | 6 months
  Pregnancy rate, cumulative pregnancy rate and ectopic pregnancy rate in order to evaluate de usefulness of the CAT test as a predictor of tubal pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Spain